CLINICAL TRIAL: NCT07292129
Title: Smartphone Addiction as a Modifiable Factor in Cervicogenic Headache: Effects on Pain, Function, Mood, and Sleep
Brief Title: Smartphone Addiction in Cervicogenic Headache
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 2025-GOKAEK-2512_2025.06.18_50
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cervicogenic Headache; Smartphone Addiction
Keywords: Headache Impact; Neck Disability; Anxiety and Depression; Sleep Disturbance; Quality of Life; Smartphone Use
MeSH Terms: conditions — Post-Traumatic Headache; Internet Addiction Disorder; Anxiety Disorders; Depression; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervicogenic Headache Group: Adults between 18 and 65 years of age diagnosed with cervicogenic headache based on the International Classification of Headache Disorders, third edition were eligible for inclusion. Exclusion criteria included systemic diseases such as diabetes mellitus, thyroid disorders, chronic kidney disease, malignancy, neurological conditions associated with neuropathic pain, and rheumatic diseases including rheumatoid arthritis, ankylosing spondylitis, or fibromyalgia. Participants with communication difficulties, illiteracy, or those who declined participation were also excluded.
- Healthy Control Group: Age- and sex-matched adults without cervicogenic headache or other chronic medical conditions served as controls. Controls were between 18 and 65 years of age, cognitively intact, literate, and willing to participate. Exclusion criteria were the same as for the cervicogenic headache group, including systemic, neurological, or rheumatological diseases, illiteracy, or refusal to participate.

SUMMARY:
Cervicogenic headache is a secondary headache disorder that originates from the cervical spine and often presents with pain radiating from the neck to the head, reduced functional capacity, and impaired quality of life. In modern society, prolonged smartphone use and dependence are increasingly recognized as potential contributors to musculoskeletal problems, poor posture, psychological distress, and sleep disturbances.

This study was designed as a case-control investigation to explore the relationship between smartphone addiction (problematic smartphone use) and clinical characteristics of cervicogenic headache in comparison with healthy individuals. Participants were evaluated in the outpatient clinics of Physical Medicine and Rehabilitation and Neurology at Yozgat Bozok University.

A structured sociodemographic form was administered, and each participant completed a set of validated assessment tools. Smartphone use behavior was assessed with the Smartphone Addiction Scale-Short Form. Headache-related disability was measured with the Headache Impact Test. Cervical function was evaluated with the Neck Disability Index. Psychological status was assessed using the Hospital Anxiety and Depression Scale. Sleep quality was examined with the Jenkins Sleep Scale. Health-related quality of life was measured using the 12-item Short Form Health Survey, and pain intensity was evaluated with the Visual Analog Scale.

The study was conducted in accordance with the Declaration of Helsinki. Approval was obtained from the Clinical Research Ethics Committee, and written informed consent was provided by all participants prior to enrollment.

DETAILED DESCRIPTION:
Cervicogenic headache is a secondary headache that arises from dysfunction or pathology of the cervical spine and associated structures. It is characterized by unilateral head and neck pain, which may radiate to the frontal or temporal regions and is often aggravated by neck movements. Cervicogenic headache is known to cause substantial functional disability, emotional distress, and reduced quality of life.

With the rapid increase in smartphone use worldwide, attention has been drawn to its possible musculoskeletal and psychological consequences. Prolonged forward head posture, repetitive neck movements, and excessive screen time may contribute to cervical dysfunction and exacerbate symptoms of cervicogenic headache. In addition, behavioral dependence on smartphones has been associated with mood disorders, sleep disturbances, and impaired daily functioning. Understanding the potential role of smartphone addiction as a modifiable factor in cervicogenic headache is therefore of clinical importance.

The present study was designed as a case-control observational protocol to investigate the association between smartphone addiction and clinical outcomes in individuals with cervicogenic headache compared with healthy controls. Data were collected in the outpatient clinics of Physical Medicine and Rehabilitation and Neurology at Yozgat Bozok University.

A standardized sociodemographic form was administered, followed by a comprehensive set of validated assessment instruments. These included the Smartphone Addiction Scale-Short Form to evaluate problematic smartphone use, the Headache Impact Test to measure the burden of headaches on daily life, the Neck Disability Index to assess functional limitations related to cervical spine disorders, the Hospital Anxiety and Depression Scale to screen for symptoms of anxiety and depression, the Jenkins Sleep Scale to evaluate sleep quality and disturbances, the 12-item Short Form Health Survey to assess physical and mental aspects of health-related quality of life, and the Visual Analog Scale to record the intensity of pain.

All assessments were performed face-to-face by trained professionals in a clinical setting. The study protocol was approved by the Clinical Research Ethics Committee. Written informed consent was obtained from each participant before enrollment, and all procedures were carried out in accordance with the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years

Literate and cognitively capable of completing questionnaires

Willing to participate and provide written informed consent

For the patient group: Diagnosis of cervicogenic headache based on the International Classification of Headache Disorders, third edition, confirmed by a neurologist

For the control group: Healthy volunteers with no known medical conditions or active complaints, age- and sex-matched with patients

Exclusion Criteria:

Comorbidities that may affect pain perception or mood, including diabetes mellitus, thyroid dysfunction, malignancy, chronic kidney disease, neurological diseases associated with neuropathic pain, rheumatoid arthritis, ankylosing spondylitis, or fibromyalgia

Illiteracy or impaired communication

Current use of medications that may interfere with outcome measures

Withdrawal of consent at any stage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cervicogenic headache according to the International Classification of Headache Disorders, third edition, confirmed by a neurologist, were recruited from the outpatient clinics of the Departments of Physical Medicine and Rehabilitation and Neurology at Yozgat Bozok University. Age- and sex-matched healthy volunteers were recruited from the same community.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale - Short Form | At baseline
  Ten-item self-report questionnaire scored on a six-point Likert scale ranging from 1 to 6. The total score ranges from 10 to 60, with higher scores indicating a greater risk of smartphone addiction. Sex-specific cut-off values are 31 or higher for males and 33 or higher for females. A Turkish validated version is available.

SECONDARY OUTCOMES:
Headache Impact Test with 6 items | At baseline
  Patient-reported questionnaire assessing the impact of headache on pain, vitality, role limitations, and emotional function. Each of the six items is scored from 6 to 13, producing a total score between 36 and 78. Higher scores indicate a greater negative impact of headache. A Turkish validated version is available.
Neck Disability Index | At baseline
  Self-reported questionnaire with ten items scored from 0 to 5. The total score is converted into a percentage ranging from 0 to 100 percent. Higher percentages indicate greater disability related to neck pain. A Turkish validated version is available.
Hospital Anxiety and Depression Scale | At baseline
  Fourteen-item questionnaire with two subscales assessing anxiety and depression, each scored from 0 to 21. Higher scores indicate more severe symptoms. Cut-off scores are defined as 0 to 7 for normal, 8 to 10 for mild, 11 to 14 for moderate, and 15 to 21 for severe symptoms. A Turkish validated version is available.
Jenkins Sleep Scale | At baseline
  Four-item questionnaire assessing sleep quality and sleep disturbances. The total score ranges from 0 to 20, with higher scores indicating poorer sleep quality. A score greater than 15 indicates clinically relevant poor sleep. A Turkish validated version is available.
Short Form-12 Health Survey | At baseline
  Twelve-item questionnaire assessing physical and mental components of health-related quality of life. It provides physical and mental component scores scaled from 0 to 100, with higher scores indicating better perceived quality of life. A Turkish validated version is available

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Demir Karakılıç, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected for this study, including questionnaire scores and demographic variables, will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The datasets will be available beginning 6 months after publication of the study results and will remain accessible for 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound proposal may request access to the de-identified datasets. Data will be shared after approval of the proposal and signing of a data access agreement. Requests should be directed to the corresponding author via the institutional email address.
URL: https://hastane.bozok.edu.tr/

REFERENCES:
- [Background] Soylu C, Kutuk B. Reliability and Validity of the Turkish Version of SF-12 Health Survey. Turk Psikiyatri Derg. 2022 Summer;33(2):108-117. doi: 10.5080/u25700. English, Turkish. PMID 35730511
- [Background] NOYAN, C.O., et al., Akıllı Telefon Bağımlılığı Ölçeğinin Kısa Formunun üniversite öğrencilerindeTürkçe geçerlilik ve güvenilirlik çalışması. Anatolian Journal of Psychiatry/Anadolu Psikiyatri Dergisi, 2015. 16.
- [Background] Aydemir, O., Hastane anksiyete ve depresyon olcegi Turkce formunun gecerlilik ve guvenilirligi. Turk Psikiyatri Derg., 1997. 8: p. 187-280.
- [Background] Telci EA, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagli N. The cultural adaptation, reliability, and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1732-5. doi: 10.1097/BRS.0b013e3181ac9055. PMID 19770615
- [Background] Dikmen PY, Bozdag M, Gunes M, Kosak S, Tasdelen B, Uluduz D, Ozge A. Reliability and Validity of Turkish Version of Headache Impact Test (HIT-6) in Patients with Migraine. Noro Psikiyatr Ars. 2020 Apr 24;58(4):300-307. doi: 10.29399/npa.24956. eCollection 2021. PMID 34924791
- [Result] Duruoz MT, Erdem D, Gencer K, Ulutatar F, Baklacioglu HS. Validity and reliability of the Turkish version of the Jenkins Sleep Scale in psoriatic arthritis. Rheumatol Int. 2018 Feb;38(2):261-265. doi: 10.1007/s00296-017-3911-2. Epub 2017 Dec 18. PMID 29250729